CLINICAL TRIAL: NCT07021807
Title: Assessing SARS-CoV-2 (COVID-19) Seroprevalence During Routine Antenatal Care Visits in Zambia
Brief Title: ANC COVID-19 Surveillance
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Other Study IDs: ANC COVID-19 Surveillance; NU2GGH002251 (Other Grant/Funding Number: Center for Disease Control and Prevention)
Record Dates: First submitted 2025-03-11; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2 Seroprevalence
Keywords: Prenatal care; Covid-19; SARS-CoV-2; sentinel surveillance; seroprevalence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to determine the seroprevalence of SARS-CoV-2 antibodies in the community with pregnant women aged 15-49 years attending first antenatal care as the sentinel population. Further, the study seeks:

* To determine the feasibility and acceptability of SARS-CoV-2 antibody tests among pregnant women
* To estimate the prevalence of HIV-COVID 19 co-infection among pregnant women aged 15-49 years
* To determine sociodemographic factors associated with SARS-CoV-2 seropositivity among pregnant women
* To compare trends in seroprevalence among pregnant women with routine surveillance data to determine if ANC sentinel surveillance is a viable surveillance strategy for SARS-CoV-2

The main question it aims to answer is:

- What is the seroprevalence of antibodies to SARS-CoV-2 among pregnant women attending first ANC visit in Zambia?

Participants will be expected to give consent to participating in the study on the day of their first antenatal visit. They should allow the collection of a dried blood spot for SARS-CoV-2 antibody test.

DETAILED DESCRIPTION:
This surveillance platform may be able to provide key information on the spread of the SARS-CoV-2 virus through the general population. By using serologic testing to understand trends in the proportion of pregnant women over time who were exposed to SARS-CoV-2, we will be able to understand not only the ultimate proportion of pregnant women who were ever infected, but also be able to track and potentially detect outbreaks (e.g. in areas with increasing positivity rates), unlike data that would be available from a single cross-sectional survey, which could give the overall prevalence at a single point in time.

Zambia is experiencing a SARS-CoV-2 epidemic. From March 18, 2020 to February 19, 2021, at total of 73,203 confirmed cases have been reported in Zambia. However, the true number is likely much larger, because surveillance systems for SARS-CoV-2 in Zambia are incomplete.

Since 2020, the coronavirus disease has become a major public health concern and sustainable and efficient surveillance platforms are urgently needed; assessing women attending 1st ANC should provide insights into transmission trends in the general population. This activity will determine what proportion of pregnant women demonstrate evidence of SARS-CoV-2 infection over time. The findings of this research may be used to change the way health system monitors the epidemic and ensures health services are made available with minimal disruptions.

The study was implemented at 39 public health facilities. A sample of 20 pregnant women attending their first ANC visit at the selected study sites will be enrolled into the study until the monthly sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnant and are registered for their first ANC visit
* Aged 15 to 49 years
* Able to provide consent to participate and have blood sample collected for the SARS-CoV-2 antibody test

Exclusion Criteria:

* Not first ANC visit for the pregnant woman
* Women less than 15 years or above 49 years old
* Women not able to provide consent for study participation

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females who are pregnant and registered for antenatal care.
Study Population: A sample of 20 pregnant women attending their first ANC visit at 39 study sites will be enrolled in the study until the monthly sample size is reached.
Sampling Method: Probability Sample
Enrollment: 9111 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 seroprevalence | 13 months
  Number of participants with a positive test result divided by the total number of participants with a valid test result by month and district.

SECONDARY OUTCOMES:
Vaccine Uptake | 13 months
  Number of participants reporting prior confirmed COVID-19 and having received a COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Oran DP, Topol EJ. Prevalence of Asymptomatic SARS-CoV-2 Infection : A Narrative Review. Ann Intern Med. 2020 Sep 1;173(5):362-367. doi: 10.7326/M20-3012. Epub 2020 Jun 3. PMID 32491919

DOCUMENTS (2):
  • Study Protocol (2021-06-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT07021807/Prot_000.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT07021807/ICF_001.pdf